CLINICAL TRIAL: NCT04484038
Title: Multicenter Study of Hypofractionated Postoperative Radiotherapy in Patients Diagnosed With Prostate Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grupo de Investigación Clínica en Oncología Radioterapia (Other)
Responsible Party: Principal Investigator, Asunción Hervas, MD, Grupo de Investigación Clínica en Oncología Radioterapia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYPORT-ES
Record Dates: First submitted 2020-07-15; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Prostate Cancer
Keywords: Radiotherapy, prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a non-randomized prospective multicenter study of hypofractionated postoperative radiotherapy in patients diagnosed with prostate carcinoma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMRT, any mode (Other): External radiation therapy with 6-18 MV photons on the 62.5 Gy prostate bed in 25 2.5 Gy fractions (EQD2 71 Gy).
  Serving per fraction: 2.5 Gy Total fractions: 25 No. fractions / week: 5 Total treatment time: 5 weeks Total nominal dose: 62.5 Gy EQD3 (TRT): 68.75 Gy EQD1.5 (CaP): 71.43 Gy EQD2 (CaP): 68.75 Gy EQD10 (TRA): 65.10 Gy
  Interventions: Radiation: hypofractionated postoperative radiation therapy

INTERVENTIONS:
Radiation: hypofractionated postoperative radiation therapy — The patients included in the study will undergo intensity-modulated radiotherapy, of any modality, and image-guided (IGRT) with an emphasis on tissue preservation and administration precision through the use of devices that guarantee the stability and reproducibility of the same.

SUMMARY:
The objective of this study is to evaluate, in patients diagnosed with prostate cancer who undergo radical prostatectomy and who require postoperative radiotherapy, tolerance in terms of acute and chronic GU and GI toxicity and efficacy in terms of biochemical control and survival, as well as of quality of life, from a hypofractional external radiotherapy scheme, increasing the dose per fraction in a shorter period of time.

DETAILED DESCRIPTION:
What the investigators present in this study is a hypofractionation scheme of 62.5 Gy in 25 daily fractions of 2.5 Gy / day, which was chosen to provide a biological equivalent dose (BED) of 166.67 Gy, comparable to the 163 Gy administered with a scheme Normally divided up to 70 Gy in daily fractions of 2 Gy / day Version 2.0, March 27, 2019

(assuming an α / β ratio of 1.5 Gy for prostate cancer). The BED in risk organs (mainly rectum and bladder) will be governed by the ratio used and will differ depending on whether acute or late toxicity is calculated. If selected an acute α / β of 10 Gy and a conservative α / β for late toxicity of 3 Gy, the standard fractionation will result in an acute BED of 84 Gy versus 78 Gy in the hypofractionation scheme and a BED of 116.67 vs. 114.5 Gy for late toxicity.

Therefore, what the investigators expect is a toxicity profile that is at least similar, if not slightly better, compared to the norm-fractionated scheme of 70 Gy in 35 fractions and similar rates of biochemical control and survival.

To all this is added the use of intensity modulated radiotherapy and image-guided radiotherapy techniques (IGRT) that will allow the investigators to significantly reduce the dose administered to risk organs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* ECOG 0-1 status.
* Previous radical prostatectomy (any modality will be allowed) with or without lymphadenectomy.
* Histological confirmation of prostate adenocarcinoma in the prostatectomy specimen.
* pT2-T3 Version 2.0, March 27, 2019
* pN0-Nx
* Indication of postoperative RT:

  * Adjuvant RT: pT3 and / or positive margins with PSA <0.2 ng / ml. Delayed RT is considered (> 6 months from the date of surgery but PSA <0.2 ng / ml).
  * Rescue RT: exclusive biochemical recurrence, without evidence of macroscopic local, regional or distant disease, after surgery. Biochemical recurrence is considered PSA ≥ 0.2 ng / ml after undetectable levels, confirmed with a subsequent determination.
* PSA levels ≤ 2 ng / ml after, at least 45 days after surgery and 30 days before inclusion in the study.
* No clinical evidence of lymph node disease. The presence will be admitted by imaging tests of pelvic nodes ≤ 1 cm in its shortest axis.
* No evidence of disease in the prostatic fossa. If you doubt by digital rectal examination or CT, an MRI will be performed.
* No evidence of distant disease after performing a thoraco-abdominal-pelvic CT scan and bone scan.
* Reasonable follow-up possibilities.
* Ability to complete the EPIC-26 questionnaire.
* Written informed consent prior to inclusion in the study.

Exclusion Criteria:

* - Previous pelvic radiation therapy.
* Distant metastasis.
* Macroscopic residual tumor.
* PSA> 2 ng / ml.
* Pathological stage T4.
* Lymph node involvement.
* Pelvic or para-aortic nodules in the reevaluation images after surgery, except pelvic nodes ≤ 1 cm in their shortest axis.
* Indication of pelvic nodal RT. Version 2.0, March 27, 2019
* Severe urinary incontinence at the time of indication for radiotherapy.
* Uni / bilateral hip prosthesis
* Previous tumors, except non-melanoma skin carcinoma, and which are not free of disease for at least 3 years from the end of the treatment of said neoplasms. Bladder tumors are excluded in all cases.
* Genetic hyper-radio-sensitivity syndromes.
* Chronic inflammatory bowel disease or partial or radical cystectomy for any reason.
* Previously treated with androgen deprivation therapy for a period greater than 3 months.
* Previously treated with chemotherapy for prostate cancer.
* Life expectancy <5 years or severe comorbidity: unstable angina, congestive heart failure, transmural myocardial infarction requiring admission in the last 6 months, active infectious process, respiratory disease requiring hospitalization, liver failure (Child-Pugh Class B or C), HIV with a CD4 count <200 cells / ml, kidney failure requiring dialysis and immunosuppressed by other causes.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-03-09 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related gastrointestinal and genitourinary acute adverse events | ≤90 days
  using the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 scale. The grades of severity from I (minimum) to V (maximum).
Incidence of late gastrointestinal and genitourinary adverse events | up to 3 years
  using the Radiation Therapy Oncology Group (RTOG) scale. The grades of severity from 1 (minimum) to 4 (maximum).

SECONDARY OUTCOMES:
Biochemical failure-free survival | up to 3 years
  Time elapsed between the date of inclusion in the study and biochemical failure
Disease-free survival (locoregional and / or remote) | up to 3 years
  Time elapsed between the date of inclusion in the study and the detection of the disease locally, regionally and / or remotely
Overall survival | up to 3 years
  Time elapsed between the date of inclusion in the study and the patient's death from any cause
Cause-specific survival | up to 3 years
  Time elapsed between the date of inclusion in the study and the patient's death due to prostate cancer or toxicity derived from treatment
Assessment of quality of life for cancer Prostate patients | at the start of treatment at 3, 12, 24 and 36 months from the end of treatment
  Use of Expanded Prostate Cancer Index questionnaire (EPIC) 26

CONTACTS AND LOCATIONS:
Overall Officials: ASUNCION R HERVAS, I, Principal Investigator — Ramon y Cajal University Hospital
Locations (19):
- Spain (19):
  - Hospital General Gregorio Marañón, Madrid, Adrid
  - Hospital Universitario de San Juan, San Juan, Alicante
  - ICO Badalona, Badalona, Barcelona
  - Hospital Dr. Negrin, Las Palmas de Gran Canaria, Gran Canaria
  - Hospital Universitario de Santiago, Santiago de Compostela, La Coruña
  - Hospital de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Torrecárdenas, Almería
  - Hospital Universitario de Badajoz, Badajoz
  - H. Sta. Cruz y San Pablo, Barcelona
  - Instituto Oncológico IMQ, Bilbao
  - Hospital Universitario San Cecilio, Granada
  - Hospital Universitario Ramón Y Cajal, Madrid
  - Fundación Jimenez Díaz 1, Madrid
  - Fundación Jiménez Díaz 2, Madrid
  - Hospital de La Princesa, Madrid
  - Hospital La Luz, Madrid
  - Hospital Quirón, Madrid
  - Hospital Ruber Internacional, Madrid
  - Complejo Hospitalario de Navarra, Pamplona

IPD SHARING:
Plan to Share IPD: No